CLINICAL TRIAL: NCT01677013
Title: Efficacy of Autologous Bone Marrow Mononuclear Cell Transplantation in Treating Selective Type 2 Diabetes Mellitus
Brief Title: Autologous Bone Marrow Mononuclear Cell Transplantation in Treating Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Lei Lei, MD, Endocrinologist, Peking University Aerospace Center Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUACH-721002
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2; diabetes mellitus; stem cell; safety; efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Oral medication treatment (No Intervention): type 2 diabetics with only oral medications
- Oral medication plus BMMCT (Experimental): Collect mononuclear cells from bone marrow aspiration, administer to pancreas via selective catheterization to splenic artery.
  Interventions: Other: BMMCT
- Oral medication plus insulin treatment (No Intervention): Type 2 diabetics who need insulin therapy with oral medications
- Oral medication plus insulin plus BMMCT (Experimental): Collect mononuclear cells from bone marrow aspiration, administer to pancreas via selective catheterization to splenic artery.
  Interventions: Other: BMMCT

INTERVENTIONS:
Other: BMMCT — Bone marrow mononuclear cell transplantation via selective catheterization
  Other Names: Bone marrow mononuclear cell transplantation
  Arms: Oral medication plus BMMCT; Oral medication plus insulin plus BMMCT

SUMMARY:
The study is aimed to evaluate the safety and efficiency of autologous bone marrow mononuclear cell transplantation in treating selective patients with type 2 Diabetes Mellitus. We hypothesized that autologous bone marrow stem cell transplantation would promote β-cells regeneration by directly differentiated from the transplanted BMMCs or stimulate local stem cells regeneration and thus decrease or eliminate the need of exogenous insulin and improve β-cells function.

DETAILED DESCRIPTION:
To study the safety and efficacy of bone marrow mononuclear cell transplantation in type 2 diabetics. According to the intervention and baseline characteristics, patients are divided into 4 arms.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* age 30-70
* stable doses of medication for at least 3 months
* BMI <35 and >18.5

Exclusion Criteria:

* secondary cause for hyperglycemia
* pregnancy or nursing
* positive autoimmune antibody of diabetes
* severe complication or concurrent diseases
* active infection or febrile illness
* allergy to iodine
* history or signs of aortic aneurysm
* history or active pancreatic diseases
* known substance abuse or alcoholism or heavy smoking
* not suitable for other conditions upon investigators' expertise

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1026 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
C-peptide | 1 year

SECONDARY OUTCOMES:
reduction of medication | 1 year
HbA1c | 1 year
adverse event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yizhong Wang, M.D., Ph.D., Study Chair — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Yuanjie Mao, M.D., Ph.D., Study Director — Department of Biochemisty, National Cerebral and Cardiovascular Center; Department of Cardiology, China-Japan Friendship Hospital; Lei Lei, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Danping Meng, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Xiyang Zhang, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Xiaolin Jia, M.D., Study Director — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Qiuming Jiang, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Yufang Li, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Song Dong, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Liyan Yang, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Hong Wang, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Mingchao Ding, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Liqin Cui, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Bin Wang, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Xin Lin, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital; Han Shi, M.D., Principal Investigator — Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital
Locations (1):
- Division of Hematology and Endocrinology, Peking University Aerospace Centre Hospital, Beijing, Beijing Municipality, China